CLINICAL TRIAL: NCT03797417
Title: The Gut Microbiome and Metabolic Activity in Patients With Vitiligo
Brief Title: Gut Microbiome and Metabolic Pathways Changes in Vitiligo
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Li Chunying-1, Vice Chief, Xijing Hospital
Other Study IDs: XJPF-LCY-V201812
Record Dates: First submitted 2019-01-05; First posted 2019-01-09 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Gut Microbiome
Keywords: Gut Microbiome; Vitiligo; Metabolic Pathways
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — the fecal and blood sample of recruited patients and healthy control volunteers
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Disease: patients with vitiligo
- Healthy Control: healthy control

SUMMARY:
Vitiligo is a chronic depigmenting autoimmune-associated skin disease and a growing psychological health concern because of its low quality of life. Genetics, immunology and environment triggers contribute to the pathophysiology of vitiligo. Identify and decrease the risk factors of vitiligo is very crucial for vitiligo treatment and prevention. Emerging evidence has linked gut microbiome to human autoimmune diseases. Here the investigators will analyze 10,913 metagenomes in stool samples from 100 adult vitiligo patients and gut microbiome associated metabolites in patients serum.

DETAILED DESCRIPTION:
Vitiligo, an autoimmune disease of the skin, is a commonly acquired chronic depigmenting disorder characterized by loss of epidermal melanocytes and progressive depigmentation clinically, affecting from 0.5% to 1% of the world population and about 1% in China Vitiligo can be a psychologically crushing associated with low quality of life, especially in colored skinned individuals. The pathoetiology of vitiligo is multifactorial and has genetic, immunological, and environmental components. Several environment-associated mechanisms have been implicated to explain melanocyte disappearance, including ultraviolet (UV) radiation exposure, repeated mechanical or thermal stress, and exposure to chemicals (especially phenols or catechols), but epidemiologic data remain limited.

Broader gut dysbioses have been identified as potential causes or contributing factors to human autoimmune diseases; however, human studies have not yet identified microbial compositional or functional triggers that are predictive of skin autoimmunity or vitiligo. Metabolites from intestinal microbiota are key determinants of host-microbe mutualism and, consequently, the health or disease of the intestinal tract. However, whether such host-microbe crosstalk influences inflammation in peripheral tissues, such as the skin, is poorly understood.

The investigators will perform a metagenome association study and serum metabolomics profiling in a cohort of vitiligo Chinese individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who volunteered and signed Informed Consent Form；
2. Male or female subjects 3-65 years of age；
3. Clinically confirmed the diagnosis of advanced vitiligo as per the diagnostic criteria for vitiligo specified in Clinical Dermatology;
4. Stable vital signs.

Exclusion Criteria:

1. Patients who had taken systemic or local treatment with vitiligo in the last month;
2. Patients who had taken systemic antibiotics，systemic hormones，cytokines, immunosuppressors in the previous three months;
3. The combination of other autoimmune diseases，gastrointestinal diseases, hepatic diseases, psychiatric and psycho-related diseases, or other skin diseases;
4. The combination of Serious, life-threatening condition such as cardiac diseases, renal diseases, endocrine system disease, cancer, or immunodeficiency diseases;
5. Women of child-bearing potential who are pregnant, plan to become pregnant during the study or are lactating；
6. Any other condition that the investigator deems unsuitable for entering the study.

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We recruit patients who have clinically advanced vitiligo, and barely have other diseases which may disturb our study results.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-09-18 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Gut microbiota sequencing results by analyzing metagenomes of 16s rRNA gene or microbial genes | 2018.10.1--2019.3.1
  Fecal samples are obtained from all recruited subjects for metagenomic sequencing. The individuals have not received any antibiotic treatment for at least one month before sample collection. In the seven days before sample collection, subjects did not take any food containing probiotics such as yogurt. Each sample was either frozen immediately at -80 °C or briefly stored in personal -20 °C freezers before transport to the laboratory within 24 h. After extracting DNA from fecal samoles, gut microbiota sequencing results by using Shotgun Strategy or Meta 16s high-throughput sequencing.
Gut microbiota associated metabolic pathways by using metabolomics profiling of serum samples study | 2018.12.1--2019.3.1
  All serum samples will be thawed on ice and a quality control (QC) sample, made by mixing and blending equal volumes (10 μl) of each serum sample, is used to estimate a mean profile representing all the analytes encountered during analysis. The acquired MS data pretreatments included peak selection and grouping, retention time correction, second peak grouping, and isotopes and adducts annotation, will be performed as previously described56. LC-MS raw data files will be converted into mzXML format and then analyzed by the XCMS and CAMERA toolbox with R statistical language.
Vitiligo associated activity measurements like VASI assays, serum markers detection | 2019.1--2019.3.1
  VASI assays will be used to evaluate patients disease condition. VASI Scoring Criteria VASI=Σall body sites (hand units) × depigmentation. Serum markers like CXCL10, IL-2, and sCD25 will be detected by ELISA kits.

CONTACTS AND LOCATIONS:
Overall Officials: Chunying Li, Principal Investigator — Study Principal Investigator
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided